CLINICAL TRIAL: NCT06907810
Title: Study of Lipid Mediators in Chronic Postoperative Pain Following Breast Cancer Surgery
Brief Title: Study of Lipid Mediators in Chronic Postoperative Pain - LICP
Acronym: LICP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Collaborators: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: LICP
Record Dates: First submitted 2025-03-11; First posted 2025-04-02 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer Female; Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Blood Specimen Collection; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Chronic pain (Experimental)
  Interventions: Other: Blood sample + questionnaire
- No chronic pain (Active Comparator)
  Interventions: Other: Blood sample + questionnaire

INTERVENTIONS:
Other: Blood sample + questionnaire — * blood sample before tumor surgery and at every follow-up visit
  * questionnaire before tumor surgery and at every follow-up visit

SUMMARY:
This interventional prospective study aims firstly to investigate variations in lipid levels in blood samples and their potential relationship with the duration and/or intensity of post-operative pain. Secondly, it aims to investigate the activation of peripheral blood mononuclear cells and neutrophils in patient blood samples. The study will enrol women aged 18 years or older who have been newly diagnosed with primary invasive or non-invasive breast cancer requiring surgical removal of the tumour, with or without axillary surgery.

The main objectives of the study are To assess whether there is an association between circulating levels of lipid mediators and chronicity (> 3 months) of postoperative pain after breast cancer surgery.

To assess whether circulating levels of lipid mediators can predict chronicity of postoperative pain in breast cancer surgery.

To assess the existence of an association between resected tissue levels of lipid mediators and chronicity of postoperative pain in breast cancer surgery.

To assess whether tissue levels of lipid mediators can predict chronicity of postoperative pain in breast cancer surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women older than 18 years
* Newly diagnosed primary invasive or non-invasive breast cancer, requiring surgical excision of the tumor, with or without axillary surgery
* Able to give informed consent

Exclusion Criteria:

* Men
* Women aged less than 18 years
* Pregnant women
* History of major psychiatric disorders
* Previous breast or axillary surgery, recurrent disease or detectable metastatic disease at the time of diagnosis
* Unable to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-03-12 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Throughout the study, an average of 2 years
  Pain intensity will be evaluated using a standardized questionnaire completed by participants at each medical consultation.
Pain duration | Throughout the study, an average of 2 years
  Pain duration will be evaluated using a standardized questionnaire completed by participants at each medical consultation.
Lipid Mediator Levels in Blood | Throughout the study, an average of 2 years
  Lipid mediator levels will be quantified in blood samples by LC-MS methods

CONTACTS AND LOCATIONS:
Overall Officials: Mireille Alhouayek, PhD, Principal Investigator — Université Catholique de Louvain
Locations (1):
- Cliniques universitaires Saint-Luc (UCLouvain), Brussels, Brussels Capital, Belgium

IPD SHARING:
Plan to Share IPD: No